CLINICAL TRIAL: NCT06672211
Title: Effect of Video-Assisted Stoma Care Education Given to Patients With Stoma on Postoperative Anxiety, Adapting to Stoma and Complications: A Randomized Controlled Trial
Brief Title: Vıdeo-Assısted Stoma Care Traınıng Gıven To Patıents Wıth Stoma Adaptıng To Stoma and Complıcatıons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hatay Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Senem GÜNEŞ KARA, Wound Care Service Manager, Hatay Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Hatay Training
Record Dates: First submitted 2024-10-21; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Stoma - Ileostomy; Stoma Colostomy; Stoma; Education of Patients
Keywords: stoma; İleostomi; Colostomy; Education of Patients

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Group receiving standard stoma care training + video-supported training
  Interventions: Other: video-supported training
- control group (No Intervention): Group receiving standard stoma care training

INTERVENTIONS:
Other: video-supported training — Patients with stomas were provided with video-supported training in addition to standard stoma care training.
  Arms: Experimental group

SUMMARY:
Objective: The aim of this study is to evaluate the effects of video-assisted stoma care training given to patients with stoma on postoperative anxiety, stoma compliance and complications.

Materials and Methods: This study was conducted as a double-blind randomized controlled interventional study within the scope of a doctoral thesis between January 2021 and September 2022 at the General Surgery Clinics of Aydın Atatürk State Hospital, Aydın State Hospital and Aydın Adnan Menderes University Practice and Research Hospital with 42 patients, 21 in the intervention group (who received video-assisted stoma care training in the postoperative period) and 21 in the control group, who met the sampling criteria. In the postoperative period, patients in the intervention group were given video-assisted stoma care training, while patients in the control group were given training using plain narration and demonstration methods. During the research process, patients were visited at 3 different time periods to determine the patients' anxiety levels, evaluate their compliance with the stoma and complications, and the patient follow-up was concluded.

ELIGIBILITY:
Inclusion Criteria:

* Having a stoma
* Being over 18 years old
* Having no complications from the stoma

Exclusion Criteria:

* Having developed any complications in the stoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Scale | Pre-training 1 day and Post-training 1 day
  The State Anxiety Inventory (STAI-I) was developed by Spielberger in 1970 and its Turkish form was adapted by Öner N. et al. for validity and reliability studies. While the anxiety level is scored as "(1) never, (2) a little, (3) a lot, and (4) completely" in the STAI-I, the options in the Trait Anxiety Inventory (STAI-II) are (1) almost never, (2) sometimes, (3) a lot, and (4) almost always. The scales include "straight" and reversed statements.

SECONDARY OUTCOMES:
Adaptation Scale for Individuals with Stoma | 1 day Pre-training and Post-training 1 day
  It is a 23-item self-assessment scale developed by Simmons et al. (2009) to determine the adaptation level of individuals with ostomy to ostomy. Its validity and reliability for Turkish was performed by Karadağ et al. (2011). Ostomy Adaptation Scale consists of 4 subdimensions including acceptance (items 1, 3, 4, 6, 9, 14, 15, 19, 23), anxiety/concern (items 12, 13, 17, 20, 21), social adaptation (items 5, 7, 8, 11) and anger (items 2 and 10). In addition, 3 items (16, 18 and 22) were not included in any subdimension. Each item in the scale is evaluated on a 5-point Likert-type scale with 0-4 points (Strongly agree, Agree, Not sure, Disagree, Strongly disagree).
Pittman Ostomy Complication Severity Index | Post-training 1 week
  Pittman Ostomy Complication Severity Index (OCSI) was developed by Joyce Pittman in 2014 to assess the frequency and severity of complications developing in the early postoperative period during the follow-up period (30 days after the operation) of individuals with stoma. Its validity and reliability in Turkish were performed by Arslantaş and Karahan (2019). OCSI was found to have content validity index (CVI = 0.9), number of items (k = 0.71-1.0), and significance between the items and the total score (ICC = 0.991, P ≤ .001). The OCSI format includes a Likert-like scale with nine individual items ranging from 0 to 3 points (minimum 0, maximum 27) and a total score calculated by summing the individual items. 0 indicates that the complication is not present, and 3 indicates that the complication is severe. The complication items considered are; discharge, peristomal irritant dermatitis, pain, bleeding, stomal necrosis, stomal stenosis, retraction, mucocutaneous separation and hyperplasi

CONTACTS AND LOCATIONS:
Overall Officials: Senem GÜNEŞ KARA, Ph.D, Study Chair — Adnan Menderes Üniversity
Locations (1):
- Adnan Menderes University Health Sciences Institute, Aydin, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Consort guidelines — https://www.equator-network.org/reporting-guidelines/consort/